CLINICAL TRIAL: NCT00106509
Title: A Randomized, Double-Blind Study of GT267-004 Versus Vancomycin, and GT267-004 Versus Metronidazole, in Patients With C.Difficile - Associated Diarrhea
Brief Title: A Study of GT267-004 Versus Vancomycin and GT267-004 Versus Metronidazole in Patients With C.Difficile - Associated Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GD3-170-301
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Clostridium Enterocolitis; Pseudomembranous Colitis
Keywords: Clostridium Enterocolitis; Pseudomembranous Colitis; Clostridium difficile-associated diarrhea; C. difficile; CDAD
MeSH Terms: conditions — Enterocolitis, Pseudomembranous

INTERVENTIONS:
Drug: tolevamer potassium-sodium (GT267-004)

SUMMARY:
Approximately 520 patients will be entered into this study taking place throughout the US and Canada. This study aims to determine if an investigational drug is safe and effective for treating symptoms of C. difficile-associated diarrhea (CDAD) and lowering the risk of repeat episodes of CDAD. The investigational drug will be evaluated in comparison to current standard antibiotic treatment, so all patients will receive active medication. All study related care is provided including doctor visits, physical exams, laboratory tests and study medication. Total length of participation is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* The presence of CDAD at the time of enrollment with no other likely etiology for the diarrhea
* Less than or equal to 48 hours of treatment with metronidazole, vancomycin or other antibacterial therapy specific for CDAD
* Baseline serum potassium > 3.0 mmol (meq)/L
* Patient considered sufficiently stable clinically to likely complete a 6 week study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520
Dates: Start 2005-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhea

SECONDARY OUTCOMES:
Time to resolution of diarrhea
Recurrence rate
Number of stools
Average stool consistency
Treatment success

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (115):
- United States (84):
  - Phoenix, Arizona
  - Rogers, Arkansas
  - Burbank, California
  - Los Angeles, California
  - Modesto, California
  - Newport Beach, California
  - Sacramento, California
  - San Diego, California
  - Denver, Colorado
  - Newark, Delaware
  - Bay Pines, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - Jacksonville, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Fort Eisenhower, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Decatur, Illinois
  - Hines, Illinois
  - Maywood, Illinois
  - North Chicago, Illinois
  - Anderson, Indiana
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Muncie, Indiana
  - Clive, Iowa
  - Des Moines, Iowa
  - Dubuque, Iowa
  - Iowa City, Iowa
  - Bowling Green, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Hagerstown, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Muskegon, Michigan
  - Rochester, Minnesota
  - Ocean Springs, Mississippi
  - Everton, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Butte, Montana
  - Missoula, Montana
  - Lebanon, New Hampshire
  - Cedar Knolls, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - Trenton, New Jersey
  - Albany, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Fargo, North Dakota
  - Akron, Ohio
  - Centerville, Ohio
  - Toledo, Ohio
  - Allentown, Pennsylvania
  - Doylestown, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Rapid City, South Dakota
  - Hermitage, Tennessee
  - Houston, Texas
  - Tyler, Texas
  - Burlington, Vermont
  - Danville, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Tacoma, Washington
  - Eau Claire, Wisconsin
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
- Canada (30):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Ajax, Ontario
  - Guelph, Ontario
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Chicoutimi, Quebec
  - Green Field Park, Quebec
  - Lévis, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Hyacinthe, Quebec
  - Sainte-Foy, Quebec
  - Trois-Rivières, Quebec
  - Saskatoon, Saskatchewan
- San Juan, Puerto Rico

REFERENCES:
- [Derived] Johnson S, Louie TJ, Gerding DN, Cornely OA, Chasan-Taber S, Fitts D, Gelone SP, Broom C, Davidson DM; Polymer Alternative for CDI Treatment (PACT) investigators. Vancomycin, metronidazole, or tolevamer for Clostridium difficile infection: results from two multinational, randomized, controlled trials. Clin Infect Dis. 2014 Aug 1;59(3):345-54. doi: 10.1093/cid/ciu313. Epub 2014 May 5. PMID 24799326